CLINICAL TRIAL: NCT06042673
Title: Impact of Pomegranate Seed Oil on Postprandial Cardiovascular Disease Risk Markers in Postmenopausal Women.
Brief Title: Impact of Pomegranate Seed Oil on Postprandial Cardiovascular Disease Risk Markers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Prof, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UREC 22/11
Record Dates: First submitted 2023-09-05; First posted 2023-09-18 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Postmenopausal Women
MeSH Terms: interventions — Nano-PSO

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pomegranate seed oil (Experimental): Participants will be asked to consume breakfast (0 minute) containing pomegranate seed oil
  Interventions: Dietary Supplement: Pomegranate seed oil
- mixed vegetable oil (Placebo Comparator): Participants will be asked to consume breakfast (0 minute) containing mixed vegetable oil
  Interventions: Dietary Supplement: Mixed vegetable oil

INTERVENTIONS:
Dietary Supplement: Pomegranate seed oil — 10 g of pomegranate seed oil+40g mixed oil (palm oil/ rapeseed oil/ safflower oil (4:0.5:0.5)) will be added to the test meal for breakfast
  Arms: Pomegranate seed oil
Dietary Supplement: Mixed vegetable oil — 50g mixed oil (palm oil/ rapeseed oil/ safflower oil (4:0.5:0.5)) will be added to the test meal for breakfast
  Arms: mixed vegetable oil

SUMMARY:
Dietary fat plays a crucial role as a modifiable risk factor influencing both non-fasting lipaemia and vascular reactivity. Notably, the intake of dietary saturated fatty acids (SFAs) has been associated with adverse effects on blood lipid profiles, whereas increased consumption of unsaturated fatty acids (UFAs) has shown potential to improve lipid health. Pomegranate seed oil (PSO) stands out due to its high content of conjugated α-linolenic acids (CLnAs). However, research comparing the impact of these fatty acids on postprandial vascular function, particularly in postmenopausal women, remains limited. A cross-over, single-blind, randomised acute postprandial study will be conducted in 15 healthy postmenopausal women. Participants will be assigned to consume the test meals either a placebo (50 g of mixed fat; 4:0.5:0.5 palm oil: rapeseed oil: safflower oil) or PSO (40 g of mixed fat and 10g of PSO) in random order on 2 separate occasions, with 4-6 weeks between each study visit. The anthropometric, blood pressure, and arterial stiffness, will be taken for each study visit. Blood samples will be collected for the measurement of fasting lipids, glucose, insulin, inflammatory markers, and whole blood culture. The findings from this study will contribute to the evidence base on how consuming meals rich in PSO influence the level of blood lipids as well as other biomarkers for cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women who have been postmenopausal for at least 12 months.
* Aged 65 and under years
* Serum TAG < 2.3 mmol/l
* Body mass index (BMI) between 18-35 kg/m2
* Fasting total cholesterol < 7.5 mmol/l
* Fasting glucose concentration <7 mmol/L

Exclusion Criteria:

* Smokers
* Medical history of myocardial infarction or stroke in the past 12 months
* Diabetes (defined as fasting glucose > 7.0 mmol/l) or other endocrine disorders
* Kidney, liver, pancreas or gastrointestinal disorder
* Hypertension (blood pressure > 140/90 mmHg), cancer, medication for hyperlipidaemia (e.g. statins), hypertension or, inflammation
* Anaemia (<115 g/L haemoglobin)
* Taking any dietary supplements known to influence lipids/gut microbiota (e.g. plant stanols, fish oil, phytochemicals, natural laxatives, probiotics and prebiotics)
* Drinking in excess of 14 units of alcohol per week
* Planning on a weight-reducing regime
* Parallel participation in another dietary intervention study
* Any other unusual medical history or diet and lifestyle habits or practices that would preclude volunteers from participating in a dietary intervention and metabolic study

Max Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-07-28 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in postprandial triacylglycerol | Acute study: taken at 0 (baseline), 30, 60, 90, 120, 180, 240, 300, 360, 420, 480 minutes
  Triacylglycerol

SECONDARY OUTCOMES:
Fasting blood lipids | Acute study: taken at 0 (baseline), 30, 60, 90, 120, 180, 240, 300, 360, 420, 480 minutes
  Total cholesterol, high density lipoprotein cholesterol
Change from baseline in postprandial insulin | Acute study: taken at 0 (baseline), 30, 60, 90, 120, 180, 240, 300, 360, 420, 480 minutes
  Insulin
Change from baseline in postprandial endothelial activation | Acute study: taken at 0 (baseline),180, 300 and 420 minutes
  E-selectin, P-selectin, vascular cell adhesion molecule 1, intercellular adhesion molecule-1
Change from baseline in postprandial blood pressure | Acute study: taken at 0 (baseline), 120, 240, 360 and 480 minutes
  Systolic and diastolic blood pressure Systolic and diastolic blood pressure Systolic and diastolic blood pressure Systolic and diastolic blood pressure
Change from baseline endothelial microvascular function | Acute study: taken at 0 (baseline),180, 300 and 420 minutes
  Laser Doppler imaging (LDI) with iontophoresis

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Food and Nutritional Sciences, University of Reading, Reading, United Kingdom

REFERENCES:
- [Derived] Almoraie MM, Spencer JPE, Wagstaff C, Jackson KG. Acute Effects of a High-Fat Meal Enriched with Pomegranate Seed Oil on Postprandial Lipemia and Endothelial Function in Postmenopausal Women: A Randomized Controlled Crossover Trial. J Nutr. 2026 Jan 22:101374. doi: 10.1016/j.tjnut.2026.101374. Online ahead of print. PMID 41580088